CLINICAL TRIAL: NCT00368706
Title: A Randomized, Double-Blind, Paralleled, Active Controlled, Multi-Center Study of the Efficacy and Safety of 5mg Solifenacin Succinate Compared to Tolterodine in Patients With Overactive Bladder
Brief Title: A Double-Blind, Paralleled Study Comparing Efficacy/Safety of Solifenacin to Tolterodine in Overactive Bladder Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 90506/CHoTD01
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Urinary Bladder, Overactive
Keywords: solifenacin; Overactive bladder; Urinary incontinence; Treatment outcomes; VESIcare
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Solifenacin Succinate; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: solifenacin succinate
- 2 (Active Comparator)
  Interventions: Drug: tolterodine

INTERVENTIONS:
Drug: solifenacin succinate — Oral
  Other Names: Vesicare; YM905
  Arms: 1
Drug: tolterodine — oral
  Arms: 2

SUMMARY:
To evaluate the efficacy and safety of solifenacin succinate (Vesicare) 5mg OD in subjects with overactive bladder compared to tolterodine wmg, bid

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and able to complete the micturition diary correctly
* Patients experiencing frequency of micturition as verified in the diary
* Patients experiencing significant post void residual volume
* OAB symptoms including urinary frequency, urgency or urge incontinence for 3 months or more.

Exclusion Criteria:

* Significant post void residual volume
* Patients with indwelling catheters or practicing intermittent self- catheterization
* Known or suspected hypersensitivity to solifenacin succinate or other anticholinergics or lactose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of micturitions per 24 hours | 8 Weeks

SECONDARY OUTCOMES:
Change from baseline in mean volume voided per micturition | 8 Weeks
Change from baseline in mean number of incontinence episodes per 24 hours | 8 Weeks
Change from baseline in mean urgency frequency per 24 hours | 8 Weeks
Change from baseline in mean nocturia episodes per 24 hours | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Principal Investigator — Peking University First Hospital
Locations (4):
- China (4):
  - Beijing
  - Chongqing
  - Hangzhou
  - Shanghai